CLINICAL TRIAL: NCT02409498
Title: A Randomized Controlled Trial of Use of Pre-emptive Pudendal Nerve Block for Pelvic Reconstructive Surgery
Brief Title: Use of Pre-Emptive Pudendal Nerve Block for Pelvic Reconstructive Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Charles Ascher-Walsh, Director, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: GCO 13-1190
Record Dates: First submitted 2015-04-01; First posted 2015-04-06 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Pelvic Organ Prolapse
Keywords: pudendal nerve block; vaginal reconstructive surgery
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Bupivacaine; Sodium Chloride; Fluoridation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pudendal block (Active Comparator): preemptive pudendal nerve blockade with 10 ml of 0 .5 % Bupivacaine with epinephrine. 10 ml of Bupivacaine will be injected on either side using the pudendal nerve block tray.
  Interventions: Drug: pudendal block
- no pudendal block (Placebo Comparator): Saline
  Interventions: Drug: no pudendal block

INTERVENTIONS:
Drug: pudendal block — preemptive pudendal nerve blockade with 10 ml of 0 .5 % Bupivacaine with epinephrine.
  Other Names: Bupivicaine; Marcaine
  Arms: pudendal block
Drug: no pudendal block — preemptive pudendal nerve blockade with 10 ml of normal saline to each side
  Other Names: Saline; salt water; placebo
  Arms: no pudendal block

SUMMARY:
The purpose of this study is to determine the effectiveness of perineal pain control via injection of a local anesthetic to numb the pudendal nerve. The medication which is commonly used for this block is called marcaine. This is called a pudendal block it has been used in obstetrical and gynecologic surgeries for several decades. The goal of this study is to reduce the amount of pain medications taken post operatively after pelvic reconstructive surgery. Subjects undergoing pelvic reconstructive surgery will be recruited during the pre-op visit. Subjects will be asked about their pain level in the PACU and also asked to document their pain score days 1 and 2 post op. They will also be asked to keep a medication log for 14 days post op.

DETAILED DESCRIPTION:
Subjects will have a through physical exam with evolution of the pelvis support using the POP-Q (pelvic organ prolapse quantification) system. All subjects will need to sign informed consent pre-approved by the IRB. The subjects, surgeons, and anesthesiologist will all be blinded to the injected material. The OR Scrub nurse will given the envelope at the start of each case and asked to draw the material into a syringe. All subjects will receive general anesthesia. Subjects will be randomized to receive preemptive pudendal nerve blockade with 10 ml of 0 .5 % Bupivacaine with epinephrine or normal saline to each side. The allocation schedule is computer generated using random-numbers table concealed in opaque envelops. Once the patient receives general anesthesia she will be positioned appropriately in dorsal lithotomy with padded Allan stir ups. 10 ml of Bupivacaine will be injected on either side using the Iowa trumpet pudendal needle drive to direct and guide appropriate position. Aspiration was attempted for every injection to decrease the chance of intravascular infusion.

At the completion of the surgery the subjects will be brought to the PACU for care. Patients are assessed immediately upon arrival to the PACU. The patients are asked their pain level using the VAS pain scale/ modified surgical pain scale at hours 1 and 2 post op. All patients are given a prescription for Vicoprofen 7.5/200mg at their pre-op visit and asked to have it filled prior to their surgery. Patients have the option to go home the same day of surgery as long as their pain is well controlled and they are clinically stable for discharge. Continued pain management and pain scale assessment will be done at 4 hours, and post op day 1 and 2. A medication log will be kept for 2 weeks post op, detailing the number of pain medications taken during that period.

ELIGIBILITY:
Inclusion Criteria:

* The ability to read and understand English
* Be at least 18 years old
* Symptomatic Stage 2 prolapse

Exclusion Criteria:

* Intolerance to local anesthetics or narcotics
* History of major psychiatric disorder or chronic pain syndrome
* History of substance abuse or current narcotic use

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
VAS pain scale | up to 2 weeks

SECONDARY OUTCOMES:
post operative analgesic consumption | up to 2 weeks
adverse effect of the pudendal block | up to 2 weeks
Length of hospital stay | up to 2 weeks
Medical or surgical complications | up to 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mamta Mamik, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Katz J, Kavanagh BP, Sandler AN, Nierenberg H, Boylan JF, Friedlander M, Shaw BF. Preemptive analgesia. Clinical evidence of neuroplasticity contributing to postoperative pain. Anesthesiology. 1992 Sep;77(3):439-46. doi: 10.1097/00000542-199209000-00006. PMID 1519781
- [Background] Ke RW, Portera SG, Bagous W, Lincoln SR. A randomized, double-blinded trial of preemptive analgesia in laparoscopy. Obstet Gynecol. 1998 Dec;92(6):972-5. doi: 10.1016/s0029-7844(98)00303-2. PMID 9840560
- [Background] Schierup L, Schmidt JF, Torp Jensen A, Rye BA. Pudendal block in vaginal deliveries. Mepivacaine with and without epinephrine. Acta Obstet Gynecol Scand. 1988;67(3):195-7. doi: 10.3109/00016348809004200. PMID 3051873